CLINICAL TRIAL: NCT01079858
Title: Evaluation of FID 114657 in Dry Eye Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMA-09-61
Record Dates: First submitted 2010-03-02; First posted 2010-03-03 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-01

CONDITIONS: Meibomian Gland Dysfunction
Keywords: Meibomian Gland Dysfunction; Dry Eye
MeSH Terms: conditions — Meibomian Gland Dysfunction; Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FID 114657 (ORB Preserved Ocular Emulsion) (Experimental): ORB Preserved Ocular Emulsion dosed as needed throughout the day (PRN)
  Interventions: Other: FID 114657 (ORB Preserved Ocular Emulsion)

INTERVENTIONS:
Other: FID 114657 (ORB Preserved Ocular Emulsion) — Patients will dose as needed throughout the day (PRN) for 4 weeks.

SUMMARY:
The primary objective of this study is to assess the overall Meibomian Gland Dysfunction Subject's preference for a particular product. Dry eye symptom relief will also be evaluated based on clinical evaluation and a set of subject questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be at least 18 years of age
* must read and sign the informed consent forms (ICF)
* must agree to comply with the study requirements.
* Patients must have a best corrected visual acuity of 0.6 LogMar or better in each eye
* must report having an ocular examination in the last two years
* must be using topical ocular dry eye therapy (artificial tears or Restasis® at least 2 times per day.
* must have been diagnosed with Meibomian Gland Dysfunction / Posterior Blepharitis based on the following criteria: must have dry eye symptoms and Meibomian gland expression grade greater than 1.

Exclusion Criteria:

* Patients cannot wear contact lenses during the study and cannot have a history of hypersensitivity to any component of FID 114657.
* Patients cannot have ocular or intraocular surgery or serious ocular trauma within the past 6 months, and cannot have a history and/or current evidence of active intraocular inflammation in either eye.
* Patients cannot have punctal plugs that were placed less than or equal to 30 days prior to Visit 1, and they cannot have ocular conditions that, in the opinion of the investigator, preclude the safe administration of the test article.
* They cannot have started or changed the dose of chronic systemic medication within 7 days prior to visit 1, and must remain on a stable dosing regimen for the duration of the study.
* Patients cannot have participated in another investigational clinical or research study within 30 days of visit 1.
* Subjects cannot have a history and/or current evidence of the following: epithelial herpes simplex keratitis (dendritic keratitis); vaccinia, active or recent varicella viral disease of the cornea and/or conjunctiva; active ocular rosacea (excluding subjects enrolled with MGD (posterior blepharitis)); acute or chronic bacterial disease of the cornea and/or conjunctiva and/or eyelids; mycobacterial infection of the eye; and/or fungal diseases of the eye.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2010-02; Primary Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Preference based on subject's relief of dry eye | 5 weeks